CLINICAL TRIAL: NCT01723969
Title: Screening Platform of the EORTC for Clinical Trials in Advanced Colorectal Cancer "SPECTAcolor"
Brief Title: Screening Platform for Clinical Trials in Advanced Colorectal Cancer
Acronym: SPECTAcolor
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-40CRC; 2012-003714-14 (EudraCT Number)
Record Dates: First submitted 2012-11-05; First posted 2012-11-08 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; Advanced Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE blocks of tumour tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colo-rectal cancer: Tumour markers testing in patients with advanced or metastatic colo-rectal cancer
  Interventions: Genetic: Tumour markers testing

INTERVENTIONS:
Genetic: Tumour markers testing — Tumour markers testing in patients advanced or metastatic colo-rectal cancer.

SUMMARY:
The EORTC GastroIntestinal Tract Cancer Group and the EORTC HeadQuarters wish to set up a European screening platform for advanced colo-rectal cancer (CRC) patients. The goal of this screening platform is to provide quick access to new drugs to patients by offering a new structure for clinical trials.

Currently some of the most challenging clinical questions arise from the molecular sub-division of CRC that would theoretically allow to inhibit the specific, altered pathways in the patients.

A major problem for trials in this "personalized medicine" is that the low frequency of the different mutations requires a high effort for screening and identifying the patients.

The EORTC CRC screening platform will hopefully offer a feasible and efficient way to characterize the patients on the molecular basis of their tumors and allow to offer them rapid and preferential participation in clinical studies with new drugs targeted to their specific pathway alterations.

ELIGIBILITY:
Inclusion Criteria:

* Colo-rectal cancer (advanced or metastatic)
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Absence of patient's consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic colo-rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 668 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Tumour markers assessment | Within 1 week after patient registration
  Five basic tumour markers will be tested: Kras, nras, braf, MSI and PKI3

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Folprecht, MD, Study Chair — Universitaetsklinikum Carl Gustav Carus, Dresden, DE; Sabine Tejpar, MD, PhD, Study Chair — U.Z. Leuven - Campus Gasthuisberg, Leuven, BE; Daniela Aust, MD, Study Chair — Universitaetsklinikum Carl Gustav Carus, Dresden, DE
Locations (27):
- Belgium (5):
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Hopitaux Universitaires Bordet-Erasme - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Bank Of Cyprus Oncology Centre, Stróvolos, Cyprus
- Gustave Roussy Cancer Campus, Villejuif, France
- Germany (5):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Ludwig-Maximilians-Universitaet Muenchen - Klinikum der Universitaet Muenchen - Campus Grosshadern, München
  - Kliniken Oldenburg, Oldenburg
- University General Hospital Heraklion, Heraklion, Greece
- Italy (2):
  - IRCCS Azienda Ospedaliera Universitaria San Martino "IST" Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Seconda Universita Degli Studi Di Napoli, Napoli
- Poland (2):
  - The Great Poland Cancer Centre, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw
- I.P.O. Francisco Gentil - Centro De Lisboa, Lisbon, Portugal
- Spain (4):
  - Hospital General Vall D'Hebron, Barcelona
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
- Ostra Sjukhuset, Gothenburg, Sweden
- Switzerland (4):
  - Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Hopital du Valais - Hopital de Sion, Sion
  - UniversitaetsSpital Zurich, Zurich